CLINICAL TRIAL: NCT02293577
Title: Continuous Glucose Monitoring in Youth With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: HIC# 1409014566; K12DK094714 (NIH)
Record Dates: First submitted 2014-11-07; First posted 2014-11-18 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: continuous glucose monitor — In this study all subjects will wear a continuous glucose monitor for 5 days.

SUMMARY:
The purpose of this study is to use a continuous glucose monitor (CGM) to describe the day to day blood glucose variability in youth with type 2 diabetes. The hypothesis is that CGM will identify caloric and exercise related variation in blood glucose that is not identified by the subjects' current regimen of intermittent finger stick blood glucose measurements.

DETAILED DESCRIPTION:
The TODAY study and other studies have reported disappointing results of intensive life-style programs alone or in combination with metformin in maintaining optimal control of type 2 diabetes (T2D) in adolescents. Continuous glucose monitoring (CGM) has been successful in lifestyle modification in adults with T2D but use of CGM has not been studied in youth with T2D. Thus the feasibility of this technology should be evaluated in this patient population as it may prove to be an effective adjunct to treatment in the future.

Youth with type 2 diabetes will be approached for enrollment in this study. The study will be explained to volunteers who meet eligibility criteria and informed consent/assent will be obtained. Demographic data will be recorded. A medical history will be performed. A urine pregnancy test (in women) will be measured to confirm eligibility. Height, weight, BMI, percent body fat, fat mass, and fat free mass will be measured. Hemoglobin A1c (HbA1c) will be measured. After enrollment a blinded CGM will be placed. CGM is a device inserted under the skin on the abdomen which monitors glucose levels every 5 minutes, recording this information. CGM is commonly worn by kids with type 1 diabetes. The study will allow collection of information on glucose variability in much greater detail than can be seen from intermittent fingerstick glucose values or from an oral glucose tolerance test. Subjects will meet with a nutritionist to learn how to keep a food record. They will be given empty food records to complete for each day. They will also be given an accelerometer and instructed in its use, however they will remain blinded to the data obtained. The study will be 5 days in length. Subjects will be urged to continue their normal eating and activity behaviors. During the study period blood sugar and CGM data will be recorded via glucometer and sensor downloads, dietary intake via food record, and activity via accelerometer. Glucometer testing of blood glucose is required at least every 12 hours to calibrate the CGM. To minimize the need for overnight tests to calibrate the CGM, subjects will be asked to check their blood sugar using a glucometer 3 times a day, preferably fasting in the morning before breakfast, before dinner, and at bedtime. To optimize the accuracy of dietary intake records, subjects will be contacted frequently and the food record information recorded by study personnel. Subjects will be given a "morning checklist" to keep in a visible area to improve compliance by reminding them to keep study devices with them all day. At the follow-up visit the CGM will be downloaded revealing blood glucose tracings for the study period. Additionally the completed food records will be collected and the accelerometer will be downloaded.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 2 diabetes
* Duration of type 2 diabetes ≥ 3 months
* Naïve to continuous glucose monitoring
* Willing to wear a continuous glucose monitor for 5 days
* Willing to check blood sugar at least every 12 hours, preferably 3 times a day
* Willing to wear an accelerometer for 5 days
* Willing to keep a food record for 5 days, including frequent phone contact from the research staff
* Be in good general health without other acute or chronic illness that in the judgment of the investigator could interfere with the study or jeopardize subject safety
* Able to give informed consent (for children <18 years, permission from parents and subject assent will be required)
* Female subjects of reproductive potential must be abstinent or consistently using appropriate family planning methods

Exclusion Criteria:

* Presence of any medical or psychiatric disorder that may interfere with subject safety or study conduct
* Use of any medications (besides insulin and/or metformin) known to effect blood glucose levels, including oral or other systemic glucocorticoid therapy
* Subjects using herbal supplements will be excluded, due to the unknown effects of these supplements on glucose control
* History of hypoglycemic seizure within last year or frequent hypoglycemia (≥2 time a month)
* Female subjects who are pregnant, lactating, or unwilling to be tested for pregnancy

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Youth with type 2 diabetes will be recruited from the type 2 diabetes clinic.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2014-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Time with blood glucose >140 mg/dL | 5 days
  Subjects will be assessed for average amount of time spent with blood sugar >140, >200, and >300 mg/dL across the 5 day study period.
Glycemic excursion after caloric intake | 5 days
  Glycemic excursion after caloric intake will be assessed using the mean change (delta) blood glucose meal time to 2-4 hours afterwards over the 5 day study period.
Glucose area under the curve | 5 days
  Continuous Glucose Monitoring (CGM) glucose readings will be averaged across the 5 day period and used to obtain the area under the curve.
Average glucose | 5 days
  Continuous Glucose Monitoring (CGM) glucose readings will be used to obtain the average glucose levels for subjects across the 5 day period.
Peak glucose | 5 days
  Continuous Glucose Monitoring (CGM) glucose readings will be used to obtain the peak glucose level for subjects over the 5 day period.
Time with blood glucose >200 mg/dL | 5 days
  Subjects will be assessed for average amount of time spent with blood sugar >140, >200, and >300 mg/dL across the 5 day study period.
Time with blood glucose >300 mg/dL | 5 days
  Subjects will be assessed for average amount of time spent with blood sugar >140, >200, and >300 mg/dL across the 5 day study period.

SECONDARY OUTCOMES:
Caloric intake | 5 days
  Food diaries will be used to quantify and assess the average daily caloric intake of subjects across the 5 day study period.
Total fat intake | 5 days
  Food diaries will be used to quantify and assess the average daily caloric intake of subjects across the 5 day study period. The percent kcal from total fat will be obtained from these data.
Sugar intake | 5 days
  Food diaries will be used to quantify and assess the average daily caloric intake of subjects across the 5 day study period. The percent kcal from sugar will be obtained from these data.
Protein intake | 5 days
  Food diaries will be used to quantify and assess the average daily caloric intake of subjects across the 5 day study period. The percent kcal from protein will be obtained from these data.
Physical Activity | 5 days
  Subjects will have their average daily physical activity measured via accelerometer. The average number of "steps" is the outcome of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Van Name, Principal Investigator — Yale University
Locations (1):
- Yale Pediatric Diabetes Research Program, New Haven, Connecticut, United States